CLINICAL TRIAL: NCT02417181
Title: The (Cost-)Effectiveness of Physician Assistants Working at the Primary Out of Hours Emergency Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Kwaliteit en Ontwikkeling Huisartsenzorg (Other); GP Cooperative Emmen (CHD Emmen) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PA_in_spoedzorg
Record Dates: First submitted 2015-03-31; First posted 2015-04-15 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Primary Healthcare; Out-of-hours Medical Care
Keywords: Physician assistants; Out-of-hours medical care; Primary healthcare; Emergency Medical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Practitioners Care (No Intervention): Usual medical care provided by a general practitioner at the out-of-hours primary care service
- Physician Assistants Care (Experimental): Medical care provided by the Physician Assistant at the out-of-hours primary care service
  Interventions: Other: Care provided by Physician Assistants

INTERVENTIONS:
Other: Care provided by Physician Assistants — Patients will receive care at the out-of-hours primary care service by a Physician Assistant instead of a General Practitioner (substitution of care from physicians to nurses).
  Arms: Physician Assistants Care

SUMMARY:
The aim of this study is to explore the effect of substituting General Practitioners (GPs) by Physician Assistants (PAs) in out-of-hours primary care. Effects are measured in terms of the implication for the care model, quality of care delivered by PAs in comparison to GPs; the complaints treated by PAs in comparison to GPs; safety, efficiency and patient satisfaction. Lastly, this study will provide insight in the changes in costs of healthcare.

DETAILED DESCRIPTION:
Out-of-hours care in the Netherlands is under pressure. Workload for general practitioners (GPs) during out-of-hours care is high and there are concerns about maintaining the quality of care. Since 80% of the complaints shown in out-of-hours care are low complex and not urgent, not all patients necessarily have to be seen by a physician. Shifting care from GPs to physician assistants (PAs) is considered to be a possible method to reduce workload while maintaining high quality and safety of care.

Previous research, on PAs in primary care during office hours, has shown PAs were found to be acceptable, effective and efficient in complementing the work of GPs.

We hypothesize that in a team of PAs and GPs working out-of-hours primary care, the PAs will deliver care to less urgent and complex complaints, deliver quality of care comparable to GPs and their implementation will lead to a reduction in cost of healthcare.

We compare care provided by a team of PAs and GPs with a team of only GPs. Within the team of PAs and GPs we make a comparison between the two healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Patients (with urgency U2, U3, U4, or U5) requesting an appointment at the primary out of hours emergency service during the weekend between 9.00 and 17.00 hours.

Exclusion criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10161 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of patients | 18 months
  To measure substitution of healthcare, the number of consultations in the experimental and control group and per discipline will be measured. These data will be derived from the electronic medical records.
Patient characteristics (composite) | 18 months
  Patient characteristics of patients seen in the experimental and control group and per discipline include age, gender, urgency and type of complaint. These data will be derived from the electronic medical records.

SECONDARY OUTCOMES:
The number of prescriptions; number of test & investigations ordered and referral to the emergency department | 18 months
  The performance of the two conditions as well as the disciplines will be measures by number of prescriptions; number of test & investigations ordered and referral to the emergency department. These data will be derived from the electronic medical records.
Direct healthcare costs related to care provide by PAs and GPs will be calculated. | 18 months
  Costs related to care provided in the experimental and control group, and per discipline will be calculated, including number of consultations, resource use, referrals, and prescriptions.
Adherence to the practice guidelines for General Practitioners | 6 months
  Adherence of the PA to the practice guidelines for General Practitioners will be measured by video recordings of in total 30 consultations/visits of the PA. Two independent General Practitioners will score the adherence by a list of indicators. Outcomes will be compared by scores of GPs and Nurse Practitioners (measured in previous research).
Amount of adverse events and complications | 18 months
  The amount of adverse events and complications will be recorded, as well as complaints by the patients.
Patient satisfaction questionaire | 6 months
  Patient satisfaction will be measured using an abridgment of the CQ-index questionnaire. During the intervention period 200 questionnaires will be sent to patients who had either a consult with the PA or with the GP at the out-of-hours primary care service. Results will be compared with results on the CQ-index of the GP and NP (measured in previous research)
Knowledge test concerning frequently presented complaints | 1 month
  Knowledge of PAs will be measured with regard to a number of frequently presented complaints by using a knowledge test. Results are compared with the results on the knowledge test of GPs and NPs (measured in previous research).

CONTACTS AND LOCATIONS:
Locations (1):
- Centrale Huisartsendienst Drenthe, Emmen, Netherlands